CLINICAL TRIAL: NCT01029184
Title: Assessment of Tolerance of Cereals in Infants With Atopic Symptoms
Brief Title: Tolerance of Cereals for Atopic Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to enrol and as a pilot study sample size was not powered anyway
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07.47.INF
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Allergy
Keywords: weaning; cereals; allergy; atopy; open allergenic test
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- complete non allergenic cereals (Active Comparator): existing commercialized product
  Interventions: Other: commercialized complete cereals
- complete non allergenic cereals plus (Experimental): commercialised product with the addition of a novel ingredient
  Interventions: Other: commercialized complete cereals with additional ingredient

INTERVENTIONS:
Other: commercialized complete cereals — complete cereals suitable for the weaning period
  Arms: complete non allergenic cereals
Other: commercialized complete cereals with additional ingredient — complete cereals suitable for weaning period
  Arms: complete non allergenic cereals plus

SUMMARY:
In this study, non allergenic cereals will be tested in infants with atopic symptoms. The test will be performed in a hospital.

DETAILED DESCRIPTION:
In the majority of food allergy cases, an exclusion diet results in regression of clinical symptoms but this diet may not be nutritionally complete. To feed a baby who has a food allergy, we want a food with low allergenic ingredients.

For this reason, a complete cereal has been specially developed and formulated for the weaning period of infants and young children suffering from milk, soy or wheat protein allergy or hypersensitivity due to celiac disease.

It allows a smooth transition into and through the weaning period. The ingredients of this product are all from vegetable sources and it is therefore suitable for a vegetarian diet. It has been commercialised for many years and has proved to be completely safe, however so far no study has been specifically designed and powered to assess tolerance of this product in infants with atopic symptoms.

In this study we are testing the tolerance (symptoms stability) of non allergenic cereals during an open allergenic test in infants with atopic symptoms and/or positive Skin Prick Test (SPT) or positive specific RAST-IgE or positive Patch Test. We are also testing the same product containing an additional ingredient with a potential effect in allergy management.

Such complete cereals is a very good option for allergic children in comparison to an exclusion diet that may not be nutritionally complete.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged from 4 to 40 months at the time of enrolment
* With atopic symptoms and/or positive Skin Prick Test (SPT) or positive specific RAST-IgE or positive Patch Test
* Infants who received a specific elimination oligoallergenic diet from the study site for at least 5 days before the day of enrolment
* Having obtained his/her signed legal representative's informed consent

Exclusion Criteria:

* Infant on systemic drugs (e.g. antihistamines) according to half-life at time of enrolment
* Congenital illness or malformation that may affect normal growth (especially immunodeficiency)
* Infant whose parents / caregivers cannot be expected to comply with treatment.
* Infant currently participating in another interventional clinical trial

Ages: 4 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Documentation of atopic symptoms and clinical examination for presence or absence of some objective and subjective symptoms with evaluation of severity (SCORAD) if necessary | 48 hours

SECONDARY OUTCOMES:
Morbidity will be assessed by the frequency of adverse events | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kinderarzt-Allergologie-Sportmedizin Fachklinik Gaißach, Gaißach Bei Bad Tölz, Germany